CLINICAL TRIAL: NCT00261976
Title: Long-term Safety Follow-up of REMICADE (RESULTS)
Brief Title: A Long-term Safety Study of Infliximab (Remicade)
Status: Completed | Type: Observational
Sponsor: Centocor, Inc. (Industry)
Collaborators: Centocor BV (Industry)
Responsible Party: Sponsor
Other Study IDs: CR004780; C0168T45 (Other: Centocor, Inc)
Record Dates: First submitted 2005-12-02; First posted 2005-12-06 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Arthritis, Rheumatoid; Crohn Disease; Psoriasis
Keywords: Rheumatoid arthritis; Crohn's disease; Psoriasis
MeSH Terms: conditions — Arthritis, Rheumatoid; Crohn Disease; Psoriasis | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients in infliximab clinical studies: All patients enrolled in selected Centocor sponsored infliximab clinical studies.
  Interventions: Drug: Infliximab (Remicade)

INTERVENTIONS:
Drug: Infliximab (Remicade) — This is an non-interventional study. Participants took the study product as part of their medical routine.

SUMMARY:
This is a study evaluating the long-term safety of infliximab (Remicade)

DETAILED DESCRIPTION:
The purpose of this study is to collect long-term safety information on infliximab (Remicade) from patients who participate in research studies using those drugs. All patients in these studies are being asked to participate in this long-term safety follow-up study which will provide important information about the study drug. The long-term effect of the study drug on survival, serious infections, new malignancies and new autoimmune diseases will be measured from data collected over a 5-year period. Additional information about possible delayed allergic reactions (possible fever, rash, fatigue, joint pain) will also be collected if you received infliximab (Remicade) after the end of the primary study. Study participation in this research study is 5 years after the end of the primary study. Questionnaires will be completed about patient's health and the occurrence of these safety events at intervals of 6 months, 1 year, 2 years, 3 years, 4 years and 5 years after patients complete participation in the primary study.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled in ongoing and future Centocor sponsored infliximab clinical studies that require long-term safety follow-up (ie, primary studies). Patients must have received at least 1 dose of study agent to be eligible for participation in the study

Exclusion Criteria:

- Did not previously participate in Centocor sponsored infliximab clinical studies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients enrolled in ongoing and future Centocor sponsored infliximab clinical studies.
Sampling Method: Non-Probability Sample
Enrollment: 2971 (Actual)
Dates: Start 2002-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with each of the following long-term safety events | Five years
  Number of patients with each of the following long-term safety events: serious infections, new malignancies, new autoimmune diseases, death, or delayed hypersensitivity (serum sickness-like) reactions.

SECONDARY OUTCOMES:
Number of patients with malignancies by malignancy type | Five years
  Number of patients with malignancies by malignancy type (ie, lymphoma, nonmelanoma skin cancers, other malignancies).
Number of patients with serious infections by type of infection | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (205):
- United States (100):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Montgomery, Alabama
  - Paradise Valley, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Anaheim, California
  - Fresno, California
  - Irvine, California
  - Los Angeles, California
  - Madera, California
  - Orange, California
  - Pasadena, California
  - Rancho Mirage, California
  - San Diego, California
  - Santa Monica, California
  - Stanford, California
  - Torrance, California
  - Denver, Colorado
  - Hamden, Connecticut
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Waterbury, Connecticut
  - Aventura, Florida
  - Largo, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Alpharetta, Georgia
  - Atlanta, Georgia
  - Marietta, Georgia
  - Coeur d'Alene, Idaho
  - Chicago, Illinois
  - Evanston, Illinois
  - Gurnee, Illinois
  - Maywood, Illinois
  - Normal, Illinois
  - Rockford, Illinois
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Overland Park, Kansas
  - Wichita, Kansas
  - Louisville, Kentucky
  - Portland, Maine
  - Baltimore, Maryland
  - Greenbelt, Maryland
  - Wheaton, Maryland
  - Andover, Massachusetts
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Ann Arbor, Michigan
  - Detroti, Michigan
  - East Lansing, Michigan
  - Grand Rapids, Michigan
  - Edina, Minnesota
  - Fridley, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Reno, Nevada
  - Voorhees Township, New Jersey
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Lake Oswego, Oregon
  - Portland, Oregon
  - Bethlehem, Pennsylvania
  - Lancaster, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia Pennsylvan, Pennsylvania
  - West Reading, Pennsylvania
  - Willow Grove, Pennsylvania
  - North Charleston, South Carolina
  - Goodlettsville, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Lubbock, Texas
  - San Antonio, Texas
  - Burlington, Vermont
  - Salem, Virginia
  - Bellevue, Washington
  - Kirkland, Washington
  - Seattle, Washington
  - Spokane, Washington
  - Milwaukee, Wisconsin
- Argentina (5):
  - Buenos Aires
  - Córdoba
  - Cp
  - Rosario
  - San Miguel de Tucumán
- Austria (3):
  - Graz
  - Innsbruck
  - Vienna
- Belgium (7):
  - Brussels
  - Diepenbeek
  - Edegem
  - Genk
  - Ghent
  - Leuven
  - Liège
- Canada (26):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Richmond, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Kitchener, Ontario
  - London, Ontario
  - Markham, Ontario
  - Newmarket, Ontario
  - North Bay, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Waterloo, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec
  - Ste-Foy, Quebec
  - Halifax
  - Hamilton Ontario
  - Montreal
  - Saskatoon
- Denmark (5):
  - Aarhus
  - Hellerup
  - Hvidovre
  - København NV
  - Odense
- Finland (4):
  - Helsinki
  - Hus
  - Jyväskylä
  - Pikonlinna
- France (7):
  - Créteil
  - Montpellier
  - Nantes
  - Nice
  - Paris
  - Pierre-Bénite
  - Poitiers
- Germany (13):
  - Berlin
  - Bochum
  - Cologne
  - Dresden
  - Erlangen
  - Frankfurt
  - Hamburg
  - Leipzig
  - Mainz
  - Münster
  - Oldenburg
  - Würzburg
  - Wÿrzburg
- Hungary (2):
  - Budapest
  - Debrecen
- Dublin, Ireland
- Israel (2):
  - Haifa
  - Tel Aviv
- Netherlands (4):
  - Amsterdam-Zuidoost
  - Maastricht
  - Rotterdam
  - Utrecht
- Oslo, Norway
- Poland (6):
  - Bialystok
  - Lublin
  - Szczecin
  - Warsaw
  - Wroclaw
  - Włoszczowa
- Spain (5):
  - Barcelona
  - Buenos Aires
  - Córdoba
  - Federal
  - Madrid
- Gothenburg, Sweden
- Switzerland (2):
  - Geneva
  - Zurich
- United Kingdom (11):
  - Bath
  - Birmingham
  - Cambridge
  - Cannock
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Newcastle upon Tyne
  - Norwich
  - Oxford

REFERENCES:
- See also: Study results from the long term safety follow-up of REMICADE (RESULTS) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=150&filename=CR004780_CSR.pdf